CLINICAL TRIAL: NCT02550288
Title: A Phase III, Randomized, Active Comparator-controlled Clinical Trial to Study the Efficacy and Safety of MK-0653C in Japanese Patients With Hypercholesterolemia
Brief Title: A Clinical Trial to Assess the Efficacy and Safety of MK-0653C in Japanese Participants With Hypercholesterolemia (MK-0653C-383)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653C-383; 153060 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2015-09-14; First posted 2015-09-15 (Estimated); Results first posted 2017-06-21 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Atorvastatin; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Ezetimibe 10 mg (Active Comparator): 1 ezetimide 10 mg tablet, 2 atorvastatin 10 mg placebo capsules orally once daily for 12 weeks.
  Interventions: Drug: Ezetimibe 10 mg; Drug: Placebo for Atorvastatin 10 mg capsule; Behavioral: Diet control/Daily Exercise
- Atorvastatin 10 mg (Active Comparator): 1 atorvastatin 10 mg capsule, 1 ezetimide 10 mg placebo tablet, and 1 atorvastatin 10 mg placebo capsule orally once daily for 12 weeks.
  Interventions: Drug: Atorvastatin 10 mg; Drug: Placebo for Ezetimibe 10 mg tablet; Drug: Placebo for Atorvastatin 10 mg capsule; Behavioral: Diet control/Daily Exercise
- Atorvastatin 20 mg (Active Comparator): 2 atorvastatin 10 mg capsules and 1 ezetimide 10 mg placebo tablet orally, once daily for 12 weeks.
  Interventions: Drug: Atorvastatin 10 mg; Drug: Placebo for Ezetimibe 10 mg tablet; Behavioral: Diet control/Daily Exercise
- Ezetimibe 10 mg + Atorvastatin 10 mg (Experimental): 1 Ezetimibe 10 mg tablet, 1 atorvastatin 10 mg capsule and 1 atorvastatin 10 mg placebo capsule orally, once daily for 12 weeks
  Interventions: Drug: Ezetimibe 10 mg; Drug: Atorvastatin 10 mg; Drug: Placebo for Atorvastatin 10 mg capsule; Behavioral: Diet control/Daily Exercise
- Ezetimibe 10 mg + Atorvastatin 20 mg (Experimental): 1 Ezetimibe 10 mg tablet and 2 atorvastatin 10 mg capsules orally, once daily for 12 weeks
  Interventions: Drug: Ezetimibe 10 mg; Drug: Atorvastatin 10 mg; Behavioral: Diet control/Daily Exercise

INTERVENTIONS:
Drug: Ezetimibe 10 mg
  Arms: Ezetimibe 10 mg; Ezetimibe 10 mg + Atorvastatin 10 mg; Ezetimibe 10 mg + Atorvastatin 20 mg
Drug: Atorvastatin 10 mg
  Arms: Atorvastatin 10 mg; Atorvastatin 20 mg; Ezetimibe 10 mg + Atorvastatin 10 mg; Ezetimibe 10 mg + Atorvastatin 20 mg
Drug: Placebo for Ezetimibe 10 mg tablet
  Arms: Atorvastatin 10 mg; Atorvastatin 20 mg
Drug: Placebo for Atorvastatin 10 mg capsule
  Arms: Atorvastatin 10 mg; Ezetimibe 10 mg; Ezetimibe 10 mg + Atorvastatin 10 mg
Behavioral: Diet control/Daily Exercise — Diet and Daily exercise program as per Japan Atherosclerosis Society Guideline 2012 (JAS2012)

SUMMARY:
This study will evaluate the efficacy and safety of MK-0653C (Ezetimibe [EZ] 10 mg/Atorvastatin [Atora] 10mg or 20 mg) compared to EZ 10 mg, Atora 10 mg, or Atora 20 mg alone when administered to Japanese participants with hypercholesterolemia. The primary hypothesis is that MK-0653C (EZ 10 mg/Atorva 10 mg) is superior to EZ 10 mg and is superior to Atorva 10 mg and that MK-0653C (EZ 10 mg/Atorva 20 mg) is superior to EZ 10 mg and is superior to Atorva 20 mg in percent change from baseline in low-density lipoprotein cholesterol (LDL-C) after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Japanese outpatient with hypercholesterolemia.
* Females must be non-reproductive potential or agree to remain abstinent or use (or partner use) two acceptable methods of birth control from date of signed informed consent to the 14 days after the last dose of study drug
* Agree to maintain a stable diet that is consistent with the Japan Atherosclerosis Society Guideline 2012 (JAS2012) for prevention of atherosclerotic cardiovascular diseases for the duration of the study

Exclusion Criteria:

* Uncontrolled hypertension
* Type 1 or uncontrolled type 2 diabetes mellitus (treated or untreated)
* History of coronary artery disease (CAD) Homozygous familial hypercholesterolemia or has undergone LDL apheresis
* Had a gastrointestinal tract bypass, or other significant intestinal malabsorption
* History of cancer within the past 5 years except for successfully treated dermatological basal cell or squamous cell carcinoma or in situ cervical cancer
* Human immunodeficiency virus (HIV) positive
* History of drug/ alcohol abuse within the past 5 years or psychiatric illness not adequately controlled and stable on pharmacotherapy
* Consumes more than 25 g of alcohol per day
* Consumes more than 1L of grapefruit juice per day
* Currently following an excessive weight reduction diet
* Engaging in a vigorous exercise regimen (e.g.; marathon training, body building training etc.) or intends to start training during the study
* Hypersensitivity or intolerance to ezetimibe or atorvastatin
* History of myopathy or rhabdomyolysis with ezetimibe or any statin
* Pregnant or lactating
* Taking any other investigational drugs and/or has taken any investigational drugs within 30 days

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teramoto T, Yokote K, Nishida C, Tershakovec AM, Oshima N, Takase T, Hirano T, Lee R, Johnson-Levonas AO. A phase III, clinical trial to study the efficacy and tolerability of ezetimibe plus atorvastatin combination therapy in Japanese patients with hypercholesterolemia: a randomized, double-blind comparative study. J Clin Therapeut Med. 2017;33(7):551-567

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consisted of screening, a 2-week placebo run-in and a 12-week treatment period.
Period: Overall Study
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Started | 35 | 68 | 69 | 68 | 69
Completed | 33 | 65 | 68 | 65 | 66
Not Completed | 2 | 3 | 1 | 3 | 3
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 2 | 1 | 0 | 3
Not completed — Participant moved | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Total
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (9.8) | 58.9 (8.6) | 58.3 (10.3) | 58.7 (10.4) | 57.9 (11.0) | 58.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 34 | 39 | 34 | 37 | 162
  Male | 17 | 34 | 30 | 34 | 32 | 147

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: Participants had LDL-C levels assessed at baseline and after 12 weeks of study drug administration. The change from baseline was calculated.
Time Frame: Baseline and Week 12
Population: All participants who received at least 1 dose of study treatment, and had a baseline observation or at least 1 post-baseline observation. One participant who received misallocated study medication during placebo run-in period was excluded from the main population for the analysis of efficacy data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 68 | 68 | 69
Percentage Change | -19.3 [-22.7 to -15.8] | -44.0 [-46.5 to -41.6] | -49.1 [-51.5 to -46.7] | -55.6 [-58.0 to -53.2] | -59.2 [-61.6 to -56.8]
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Ezetimibe 10 mg + Atorvastatin 10 mg; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; Difference in Least Squares Means = -36.3, 95% CI 2-sided [-40.5 to -32.2]
Statistical Analysis 2: Comparison: Atorvastatin 10 mg vs Ezetimibe 10 mg + Atorvastatin 10 mg; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; Difference in Least Squares Means = -11.6, 95% CI 2-sided [-14.9 to -8.2]
Statistical Analysis 3: Comparison: Ezetimibe 10 mg vs Ezetimibe 10 mg + Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; Difference in Least Squares Means = -39.9, 95% CI 2-sided [-44.1 to -35.8]
Statistical Analysis 4: Comparison: Atorvastatin 20 mg vs Ezetimibe 10 mg + Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; Difference in Least Squares Means = -10.1, 95% CI 2-sided [-13.5 to -6.8]

2. Primary Outcome: Percentage of Participants Who Experience 1 or More Gastrointestinal-related Adverse Events (AEs)
Description: Gastrointestinal-related AEs included all preferred terms within system organ class of Gastrointestinal Disorders except Chapped Lips and Toothache.
Time Frame: up to 14 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 5.7 | 0.0 | 8.7 | 7.4 | 7.2

3. Primary Outcome: Percentage of Participants Who Experience 1 or More Gallbladder-related AEs
Description: Gallbladder-related AEs included Bile Duct Obstruction, Bile Duct Stone, Bile Duct Stenosis, Biliary Colic, Cholangitis, Cholecystectomy, Cholecystitis, Cholelithiasis, Gallbladder Disorder, Gallbladder Perforation, Hepatic Pain, and Hydrocholecystis.
Time Frame: up to 14 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 1.5 | 0.0 | 0.0 | 0.0

4. Primary Outcome: Percentage of Participants Who Experience 1 or More Allergic Reaction or Rash AEs
Description: Allergic Reaction or Rash AEs included Allergy to Arthropod Sting, Anaphylactoid Reaction, Anaphylactic Reaction, Anaphylatic Shock, Anaphylactoid Shock, Angioedema, Conjunctivitis Allergic, Contrast Media Reaction, Dermatitis, Dermatitis Allergic, Dermatitis Atopic, Dermatitis Bullous, Dermatitis Contact, Dermatitis Psoriasiform, Drug Hypersensitivity, Eczema, Eosinophila, Erythema, Eye Allergy, Face Oedema, Hypersensitivity, Mechanical Urticaria, Palmar Erythema, Periorbital Oedema, Photodermatosis, Photosensitivity Allergic reaction, Photosensitivity Reaction, Pigmentation Disorder, Pruritus, Pruritus Generalised, Rash, Rash Erythematous, Rash Follicular, Rash Generalised, Rash Maculo-Papular, Rash Papulosquamous, Rash Pruritic, Rash Pustular, Rash Vesicular, Rhinitis, Rhinitis Allergic, Rosacea, Skin Exfoliation, Skin Disorder, Skin Hyperpigmentation, Skin Lesion, Skin Mass, Skin Ulcer, Subcutaneous Nodule, Swelling Face, Systemic Lupus Erythematosus Rash, Urticaria.
Time Frame: up to 14 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 2.9 | 2.9 | 0.0 | 1.4

5. Primary Outcome: Percentage of Participants Who Experience 1 or More Hepatitis-related AEs
Description: Hepatitis-related AEs included Cholestasis, Cytolytic Hepatitis, Hepatic Cyst, Hepatic Failure, Hepatic Lesion, Hepatic Necrosis, Hepatitis, Hepatitis Cholestatic, Hepatitis Fulminant, Hepatitis Infectious, Hepatocellular Injury, Hepatomegaly, Jaundice, Jaundice Cholestatic.
Time Frame: up to 14 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

6. Primary Outcome: Percentage of Participants Who Experience Consecutive Elevations in Alanine Aminotransferase (ALT) ≥3 Times Upper Limit of Normal (ULN)
Description: Participants had ALT levels assessed throughout the 12 week treatment period. Participants who had 2 consecutive assessments of ALT that were 3 x ULN or greater were recorded. The ALT ULN was 40 U/L.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 0.0 | 0.0 | 1.5 | 0.0

7. Primary Outcome: Percentage of Participants Who Experience Consecutive Elevations in Aspartate Aminotransferase (AST) ≥3 Times ULN
Description: Participants had AST levels assessed throughout the 12 week treatment period. Participants who had 2 consecutive assessments of AST that were 3 x ULN or greater were recorded. The AST ULN was 40 U/L.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 0.0 | 0.0 | 1.5 | 0.0

8. Primary Outcome: Percentage of Participants Who Experience Consecutive Elevations in ALT and/or AST ≥3 Times ULN
Description: Participants had ALT and AST levels assessed throughout the 12 week treatment period. Participants who had 2 consecutive assessments of ALT and/or AST that were 3 x ULN or greater were recorded. The ALT and AST ULNs were 40 U/L.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 0.0 | 0.0 | 1.5 | 0.0

9. Primary Outcome: Percentage of Participants Who Experience Consecutive Elevations in ALT ≥5 Times ULN
Description: Participants had ALT levels assessed throughout the 12 week treatment period. Participants who had an assessment of ALT that was 5x ULN or greater were recorded. The ALT ULN was 40 U/L.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 0.0 | 0.0 | 1.5 | 0.0

10. Primary Outcome: Percentage of Participants Who Experience Consecutive Elevations in AST ≥5 Times ULN
Description: Participants had AST levels assessed throughout the 12 week treatment period. Participants who had an assessment of AST that was 5x ULN or greater were recorded. AST ULN was 40 U/L.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 69 | 69
Percentage of Participants | 0.0 | 0.0 | 0.0 | 1.5 | 0.0

11. Primary Outcome: Percentage of Participants Who Have Consecutive Elevations in ALT and/or AST ≥5 Times ULN
Description: Participants had ALT and AST levels assessed throughout the 12 week treatment period. Participants who had 2 consecutive assessments of ALT and/or AST that were 5 x ULN or greater were recorded. The ALT and AST ULNs were 40 U/L.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 0.0 | 0.0 | 1.5 | 0.0

12. Primary Outcome: Percentage of Participants Who Experience Consecutive Elevations in ALT ≥10 Times ULN
Description: Participants had ALT levels assessed throughout the 12 week treatment period. Participants who had an assessment of ALT that was 10x ULN or greater were recorded. The ALT ULN was 40 U/L.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

13. Primary Outcome: Percentage of Participants Who Experience Consecutive Elevations in AST ≥10 Times ULN
Description: Participants had AST levels assessed throughout the 12 week treatment period. Participants who had 2 consecutive assessments of AST that were 10x ULN or greater were recorded. The AST ULN was 40 U/L.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 0.0 | 0.0 | 1.5 | 0.0

14. Primary Outcome: Percentage of Participants Who Have Consecutive Elevations in ALT and/or AST ≥10 Times ULN
Description: Participants had ALT and AST levels assessed throughout the 12 week treatment period. Participants who had 2 consecutive assessments of ALT and/or AST that were 10x ULN or greater were recorded. The ALT and AST ULNs were 40 U/L.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 69 | 69
Percentage of Participants | 0.0 | 0.0 | 0.0 | 1.5 | 0.0

15. Primary Outcome: Percentage of Participants With Potential Hy's Law Condition
Description: Percentage of Participants with Potential Hy's Law Condition (defined as serum ALT or serum AST elevations >3xULN, with serum alkaline phosphatase <2xULN and total bilirubin (TBL) ≥2xULN) was summarized. The ALT and AST ULNs were 40 U/L. The ULN for alkaline phosphatase was 359 IU/L and the ULN for total bilirubin was 1.2 mg/dL.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

16. Primary Outcome: Percentage of Participants Who Have Elevations in Creatine Kinase (CK) ≥10xULN
Description: Participants had creatine phosphokinase (CK) levels assessed throughout the 12 week treatment period. Participants who had any CK level that was ≥10 x ULN were recorded. The CK ULNs for males and females were 287 IU/L and 163 IU/L, respectively.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 0.0 | 1.4 | 0.0 | 0.0

17. Primary Outcome: Percentage of Participants Who Have Elevations in CK ≥10xULN With Muscle Symptoms
Description: Participants had CK levels assessed throughout the 12 week treatment period. Participants who had any CK level that was ≥10 x ULN and had associated muscle symptoms present within +/- 7 days were recorded. The CK ULNs for males and females were 287 IU/L and 163 IU/L, respectively.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

18. Primary Outcome: Percentage of Participants Who Have Elevations in CK ≥10xULN and Drug-Related Muscle Symptoms
Description: Participants had CK levels assessed throughout the 12 week treatment period. Participants who had any CK level that was ≥10 x ULN and had associated muscle symptoms present within +/- 7 days that were reported as at least possibly-related to study drug were recorded. The CK ULNs for males and females were 287 IU/L and 163 IU/L, respectively.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of actual study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Number analyzed (Participants) | 35 | 68 | 69 | 68 | 69
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: up to 14 weeks
Arm/Group | Ezetimibe 10 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Ezetimibe 10 mg + Atorvastatin 10 mg | Ezetimibe 10 mg + Atorvastatin 20 mg
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/68 | 0/69 | 0/68 | 0/69
Other Adverse Events (participants affected / at risk) | 5/35 | 5/68 | 9/69 | 11/68 | 16/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe 10 mg (N=35) | Atorvastatin 10 mg (N=68) | Atorvastatin 20 mg (N=69) | Ezetimibe 10 mg + Atorvastatin 10 mg (N=68) | Ezetimibe 10 mg + Atorvastatin 20 mg (N=69)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe 10 mg (N=35) | Atorvastatin 10 mg (N=68) | Atorvastatin 20 mg (N=69) | Ezetimibe 10 mg + Atorvastatin 10 mg (N=68) | Ezetimibe 10 mg + Atorvastatin 20 mg (N=69)
Nasopharyngitis (Infections and infestations) | 5 (7) | 4 (4) | 8 (8) | 10 (11) | 12 (15)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.